CLINICAL TRIAL: NCT02567162
Title: Multinational Survey of Epidemiology, Morbidity, and Outcomes in Intracerebral Hemorrhage (MNEMONICH)
Brief Title: Multinational Survey of Epidemiology, Morbidity, and Outcomes in Intracerebral Hemorrhage
Acronym: MNEMONICH
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Centre for Cardiovascular Medicine and Cerebrovascular Disease Prevention (Unknown); Hospital Interzonal de Agudos San Juan Bautista (Other); Maastricht University Medical Center (Other); University of Western Ontario, Canada (Other); Northern Care Alliance NHS Foundation Trust (Other); University of Manchester (Other); University of Rostock (Other); University of Medicine and Pharmacy Craiova (Other); San Camillo de' Lellis General Hospital (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); University of Central Florida (Other); Manchester Metropolitan University (Other)
Responsible Party: Principal Investigator, Reza Behrouz, Associate Professor, The University of Texas Health Science Center at San Antonio
Other Study IDs: HSC20150655H
Record Dates: First submitted 2015-09-30; First posted 2015-10-02 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Intracerebral Hemorrhage
Keywords: Intracerebral hemorrhage; Hemorrhagic stroke; Intraparenchymal hemorrhage; Cerebrovascular disease; Stroke
MeSH Terms: conditions — Cerebral Hemorrhage; Hemorrhagic Stroke; Cerebrovascular Disorders; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this project is development of a comprehensive, prospective, multinational, multicenter, hospital-based, data repository for patients with intracerebral hemorrhage.

DETAILED DESCRIPTION:
MNEMONICH is a disease-specific registry of prospectively collected data obtained from the integration and harmonization of preexisting single-center data sets. It was formed to provide clinician-scientists around the world a comprehensive database to direct future studies toward better understanding of ICH. MNEMONICH will help examine global variability in the prevalence of ICH and identify research priorities.

New data for MNEMONICH will be prospectively collected on a wide range of features including demographics, medical history, dates and times of symptom onset, presentation symptoms, hemodynamic signs, initial and chronic medical therapy, diagnostic imaging, laboratory and genetic analyses, pathological data, and surgical and medical management. Future research will be based upon ad hoc analysis of this data.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spontaneous intracerebral hemorrhage (ICH) met by clinical and imaging criteria
* Age 18 and above
* Able to consent

Exclusion Criteria:

* ICH due to trauma
* ICH due to vascular malformation or aneurysm
* ICH due to brain tumor
* ICH due to underlying infectious lesion (e.g., abscess)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for ICH will be asked to provide their permission for the use of this information for retrospective research studies directed at ICH; such research to be conducted by the MNEMONICH investigators.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-11; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale score | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Mario Di Napoli, MD, Study Director — Centre for Cardiovascular Medicine and Cerebrovascular Disease Prevention; Mahmoud R Azarpazhooh, MD, Principal Investigator — Western University, Canada; Reza Behrouz, DO, Principal Investigator — The University of Texas Health Science Center at San Antonio; Luca Masotti, MD, Principal Investigator — Azienda USL Reggio Emilia - IRCCS; Adrian R Parry-Jones, MBChB, PhD, Principal Investigator — University of Manchester and the Salford Royal NHS Foundation Trust; Aurel Popa-Wagner, MD, PhD, Principal Investigator — University of Rostock; Mark A Slevin, PhD, Principal Investigator — Manchester Metropolitan University; Craig J Smith, MBChB, MD, Principal Investigator — University of Manchester and the Salford Royal NHS Foundation Trust; Daniel A Godoy, MD, Principal Investigator — Hospital Interzonal de Agudos San Juan Bautista; Floris H Schreuder, MD, Principal Investigator — Maastricht University Medical Center; Michael W Hoffmann, MBChB, PhD, Principal Investigator — University of Central Florida

REFERENCES:
- [Background] Behrouz R, Azarpazhooh MR, Godoy DA, Hoffmann MW, Masotti L, Parry-Jones AR, Popa-Wagner A, Schreuder FH, Slevin MA, Smith CJ, Di Napoli M; MNEMONICH Steering Committee. The Multi-National survey on Epidemiology, Morbidity, and Outcomes iN Intracerebral Haemorrhage (MNEMONICH). Int J Stroke. 2015 Dec;10(8):E86. doi: 10.1111/ijs.12629. No abstract available. PMID 26745705